CLINICAL TRIAL: NCT02503553
Title: Decision Aids in Cerebral Aneurysm Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00028774
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Cerebral Aneurysm
Keywords: option grid; neurosurgery; cerebral aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision aid (Experimental): Option grid for cerebral aneurysm treatment
  Patients will receive an option grid during the preoperative visit. They will be given the chance to ask questions. The interaction with the aneurysm surgeon will be voice recorded.
  Interventions: Behavioral: Option grid for cerebral aneurysm treatment
- Control (Placebo Comparator): Patients will receive the standard information booklet for cerebral aneurysms during the preoperative visit. They will be given the chance to ask questions. The interaction with the aneurysm surgeon will be voice recorded.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Option grid for cerebral aneurysm treatment — Patients will receive an option grid during the preoperative visit. They will be given the chance to read it and ask questions. The option grid will include head to head comparative answers for the two interventions available for cerebral aneurysms (surgical clipping and endovascular coiling). The interaction with the aneurysm surgeon will be voice recorded.
  Arms: Decision aid
Behavioral: Control — Patients will receive the standard information booklet for cerebral aneurysms during the preoperative visit. They will be given the chance to ask questions. The interaction with the aneurysm surgeon will be voice recorded.
  Arms: Control

SUMMARY:
Identifying and making a decision about the best health treatment or screening option can be difficult for patients. Decision aids can be used when there is more than one reasonable option, when no option has a clear advantage in terms of health outcomes, and when each option has benefits and harms that patients may value differently.

Decision aids may be pamphlets, videos, or web-based tools. They make the decision explicit, describe the options available, and help people to understand these options as well as their possible benefits and harms. This helps patients to consider the options from a personal view (e.g., how important the possible benefits and harms are to them) and helps them to participate with their health practitioner in making a decision.

Cerebral aneurysms are common and potentially very dangerous. However, there are important treatment choices that may prevent bleeding and stroke before aneurysm rupture.Current procedural options are clipping and endovascular coiling. The anatomy of most aneurysms is amenable to either treatment.

The treatment decisions are not simple, since each choice has its own trade-offs. How the benefits and trade-offs are valued varies across different patients, and, therefore, the right treatment decision needs to include greater patient participation. This starts with better communication of the probabilities associated with the outcomes of each option in terms that can be understood by patients. Equally important is helping the patients clarify their own treatment goals, as well as legitimizing patients' partnership in the decision-making process. Tools (e.g., decision aids) to achieve shared decision-making, are lacking in this area of medicine. We propose to investigate the impact of such decision aids on patient satisfaction and the outcomes of cerebral aneurysm coiling and clipping.

Aim 1. To determine whether structured decision aids offered to cerebral aneurysm patients are associated with increased patient participation in the decision making process as indicated by the OPTION score

Aim 2. To determine whether structured decision aids offered to cerebral aneurysm patients are associated with improved quality of life and patient satisfaction outcomes immediately preoperatively, and 30 days postoperatively.

DETAILED DESCRIPTION:
Our study will include patients presenting in the clinic with a diagnosis of cerebral aneurysm. Patients for whom surgical intervention is deemed necessary will be approached for participation in the study. After signing informed consent, they will be randomized to receive a document that will serve as a decision aid (option grid). If they are randomized as controls they will receive a standard information booklet. Patients will be given a few minutes to read through the option grid choices, and will have the chance to ask questions about the two possible treatments (cerebral aneurysm clipping, cerebral aneurysm coiling). The remainder of the interaction between patient and provider will not be affected in any other way. The physician is free to make any recommendations based on their best judgment, and the patient is free to choose based on their preferences. The visit with the patient will be voice recorded and (immediately after the completion of the encounter) will be scored based on the OPTION score, which assesses patient participation in the shared decision making process.

Patients will be interviewed again preoperatively on the day of the operation, immediately postoperatively, and 30-days postoperatively (via telephone). Performance on secondary outcome measures will be recorded.

Variables will be analyzed using Fisher exact test for categorical variables and the nonparametric Wilcoxon rank-sum test for continuous variables. Logistic regression will be performed, for each binary outcome. Linear regression will be performed for each continuous outcome.

ELIGIBILITY:
Inclusion Criteria:

* All patients for whom a decision is made to undergo cerebral aneurysm treatment

Exclusion Criteria:

* patients presenting with ruptured aneurysms/subarachnoid hemorrhage
* pediatric patients
* emergency operations with no preoperative clinic visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
OPTION score | Checked once: a) in the preoperative clinic visit
  A scale on which physician-patient interactions will be graded by an independent blinded observer (based on the voice recording) to assess patient participation in the shared-decision making process.

SECONDARY OUTCOMES:
EVAN-G | Checked once: a) within 24 hours of the operation
  A patient satisfaction score with 6 domains. The score ranges from 0-100 with higher scores representing higher satisfaction.
Change in stress level | Checked twice: a) in the preoperative clinic visit, b) immediately preoperatively on the day of the surgery
  On a scale of 0-10 with 0 being no stress and 10 being the worst stress in the patient's life.
Change in patient satisfaction level | Checked twice: a) in the preoperative clinic visit, b) immediately preoperatively on the day of the surgery
  On a scale of 0-10 with 0 being not satisfied and 10 being completely satisfied with the preoperative experience.

CONTACTS AND LOCATIONS:
Overall Officials: Kimon Bekelis, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States